CLINICAL TRIAL: NCT07390357
Title: Effect of 635-nm Photobiomodulation on Orthodontic Tooth Movement: a Randomized Split-mouth Clinical Trial
Brief Title: Effect of Photobiomodulation on Orthodontic Tooth Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Jacek Matys, Principal Investigator, Wroclaw Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WroclawMU8
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Class II Malocclusion; Orthodontic Tooth Movement
Keywords: Photobiomodulation; Orthodontics; Tooth Movement Acceleration
MeSH Terms: conditions — Overbite | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photobiomodulation-treated side (Experimental): One side of the maxilla randomly assigned to receive photobiomodulation therapy during orthodontic canine distalization. This side received standard fixed orthodontic treatment with absolute anchorage provided by orthodontic mini-implants, combined with 635-nm photobiomodulation therapy applied according to the study protocol.
  Interventions: Device: 635-nm photobiomodulation
- Sham photobiomodulation-treated side (Placebo Comparator): The contralateral side of the maxilla that served as the control. This side underwent the same orthodontic treatment protocol and mechanics as the experimental side. A sham photobiomodulation procedure was performed by placing the laser handpiece in contact with the tissues without light emission, simulating the intervention without delivering therapeutic laser energy.
  Interventions: Device: Sham photobiomodulation

INTERVENTIONS:
Device: 635-nm photobiomodulation — Photobiomodulation therapy delivered using a 635-nm diode laser in continuous wave mode. Laser irradiation was applied in contact mode to the post-extraction space and distal aspect of the canine root on the experimental side at predefined time points over a 45-day period.
  Arms: Photobiomodulation-treated side
Device: Sham photobiomodulation — A sham photobiomodulation procedure in which the laser handpiece was placed in contact with the tissues following the same schedule and application protocol as the experimental intervention, but without laser emission.
  Arms: Sham photobiomodulation-treated side

SUMMARY:
This study evaluated whether photobiomodulation (PBM), a form of low-level light therapy, can accelerate orthodontic tooth movement during canine distalization in adult patients undergoing fixed orthodontic treatment.

Eighteen adult patients requiring extraction of maxillary first premolars as part of orthodontic treatment for Class II malocclusion were enrolled. The study used a randomized, controlled, split-mouth design, in which one side of the maxilla was randomly assigned to receive PBM therapy, while the contralateral side served as an untreated control. This design allowed each participant to act as their own control.

All patients underwent standard orthodontic treatment with fixed appliances and absolute anchorage provided by orthodontic mini-implants. Canine distalization was performed using nickel-titanium closed-coil springs delivering comparable orthodontic forces on both sides. Photobiomodulation was applied on the experimental side using a 635-nm diode laser according to a predefined schedule over a 45-day period, while no laser treatment was applied on the control side.

The primary outcome was the amount of canine tooth movement, measured in millimeters at baseline and at follow-up visits using a calibrated orthodontic caliper. Tooth movement on the laser-treated side was compared with movement on the control side over time.

The purpose of this study was to determine whether photobiomodulation could safely and effectively increase the rate of orthodontic tooth movement without additional surgical intervention or pharmacological treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Class II malocclusion requiring extraction of maxillary first premolars
* Indication for maxillary canine distalization with absolute anchorage
* Fixed orthodontic treatment for the first time
* Good general health
* Non-smokers
* Good periodontal health
* Ability to understand the study procedures and provide written informed consent

Exclusion Criteria:

Uncontrolled periodontal disease

* Systemic diseases or conditions affecting bone metabolism
* Diabetes mellitus or other metabolic disorders
* Pregnancy or breastfeeding
* History of radiotherapy or bisphosphonate therapy
* Use of systemic anti-inflammatory drugs or antibiotics within the previous 12 months
* Poor oral hygiene

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
Amount of maxillary canine tooth movement | Baseline (Day 0) to Day 45
  The amount of orthodontic canine tooth movement was assessed by measuring the linear distance between the central points of the bracket slots bonded to the maxillary canine and first premolar. Measurements were performed using a calibrated orthodontic caliper at baseline (Day 0) and at follow-up visits up to Day 45. Tooth movement was calculated as the change in distance over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Ka-dent, Lipowa 18, Wschowa, Poland

IPD SHARING:
Plan to Share IPD: No